CLINICAL TRIAL: NCT02418273
Title: Denosumab for Glucocorticoid-treated Children With Rheumatic Disorders: a Pilot Study
Brief Title: Denosumab for Glucocorticoid-treated Children With Rheumatic Disorders
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: was not funded
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Erik Imel, Assistant Professor of Medicine and Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504269855
Record Dates: First submitted 2015-04-06; First posted 2015-04-16 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Osteoporosis; Juvenile Rheumatoid Arthritis; Dermatomyositis; Polyarthritis; Systemic Lupus Erythematosis; Vasculitis; Glucocorticoid-induced Osteoporosis
Keywords: denosumab; pediatric; rheumatology; osteoporosis; glucocorticoid
MeSH Terms: conditions — Osteoporosis; Arthritis, Juvenile; Dermatomyositis; Arthritis; Vasculitis | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): These subjects will receive two sequential doses of denosumab
  Interventions: Drug: denosumab
- No drug intervention (No Intervention): These subjects do not receive denosumab

INTERVENTIONS:
Drug: denosumab — These subjects will receive two doses of denosumab.
  Other Names: Prolia
  Arms: Denosumab

SUMMARY:
The purpose of this study is to evaluate denosumab as a novel treatment for bone loss in children treated with glucocorticoids for rheumatic disorders. This is a pilot Phase 1/2, randomized open-label, 12-month clinical trial of denosumab to assess its effect on bone resorption markers and bone mineral density (BMD) in children with rheumatic disorders, age 4 to 16 years, recruited within 1 month of starting a chronic systemic glucocorticoid regimen. Primary outcomes include suppression of bone turnover markers and safety assessments. Secondary outcomes include changes in bone density as measured by dual energy X-ray absorptiometry (DXA) and peripheral quantitative computed tomography (pQCT) densitometry at the radius and tibia.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate denosumab as a novel treatment for bone loss in children treated with glucocorticoids for rheumatic disorders. Children with rheumatic disorders are at risk for low bone density and fractures from the inflammatory effects of the underlying disease, and also from direct effects of glucocorticoids on bone. This is a pilot Phase 1/2, randomized open-label, 12-month clinical trial of denosumab to assess its effect on bone resorption markers and BMD in children with rheumatic disorders, age 4 to 16 years, recruited within 1 month of starting a chronic systemic glucocorticoid regimen. Two different sequential doses will be administered to the intervention group and evaluation for safety and efficacy will be conducted at study visits. Primary outcomes include suppression of bone turnover markers and safety assessments. Secondary outcomes include changes in bone density as measured by dual energy X-ray absorptiometry (DXA) and peripheral quantitative computed tomography (pQCT) densitometry at the radius and tibia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4 to 16 years of age.
2. Diagnosis of one of the following by a rheumatologist using standard criteria: juvenile dermatomyositis, juvenile idiopathic arthritis, systemic arthritis, seronegative or seropositive polyarthritis, psoriatic arthritis, systemic lupus or systemic vasculitis.
3. Within 1 month of initiating glucocorticoids ≥0.5 mg/kg prednisone equivalent daily, planned for ≥ 6 months.
4. BMD by DXA with Z-score < 0.0 on screening at lumbar spine or total body less head (TBLH).

Exclusion Criteria:

1. Previous treatment with a bisphosphonate, or other osteoporosis medication.
2. Metabolic bone disorders besides glucocorticoid-induced osteoporosis; other disorders treated with systemic glucocorticoids (inflammatory bowel disease, severe pulmonary disease, nephrotic syndrome, etc.).
3. Intent to treat with a tumor necrosis factor inhibitor or Interleukin 6 receptor antagonist during the first 6 months.
4. Glomerular filtration rate < 30ml/min [pediatric estimated glomerular filtration rate = 0.413*(height/serum creatinine)] 75
5. Planned orthopedic or other major surgery during the course of the study (at the time of enrollment)
6. Significant dental caries, or plans to undergo invasive oral procedures during the subsequent 12 months.
7. Known allergy to latex (drug packaging includes a natural rubber stopper), fructose intolerance or other denosumab contraindication.
8. 25-hydroxyvitamin D (25OHD) level < 32 ng/dl. Subjects with 25OHD <32 ng/ml may be given cholecalciferol and rescreened.
9. Hypocalcemia at screening (total serum calcium < 8.5 mg/dl after correction for albumin level).
10. Chronic ventilator dependence, or other conditions increasing risk of participation.
11. Pregnancy, or refusal to use acceptable contraception or abstain during the protocol (post-pubertal female).

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changes in bone turnover marker (N-telopeptide (NTX) /creatinine ratio). | 2 weeks, 1 month, 2 month, 3 month after each dose day.

SECONDARY OUTCOMES:
The duration of suppression of the NTX/creatinine ratio | up to six months after each dose day
The changes in bone specific alkaline phosphorus | From baseline to 1 week, 1,3,6 months after each dose day
Changes of BMD spine Z-scores | 12 month
Changes of BMD Total body less head (TBLH) Z-scores | 12 month
Changes of volumetric BMD on peripheral quantitative computed tomography | 12 month
Changes of polar strength-strain index at tibia | 12 month
Changes of polar strength-strain index at radius | 12 month
Changes in bone strength index for compression at tibia. | 12 month
Changes in bone strength index for compression at radius | 12 month
The relationships of Interleukin 6 to baseline NTX/creatinine ratio | baseline visit
The relationships of Interleukin 6 to baseline DXA | baseline visit
The relationships of Interleukin 6 to baseline pQCT variables. | baseline visit
The relationships of receptor activator of nuclear factor-kappa B ligand (RANKL) to baseline NTX/creatinine ratio | baseline visit
The relationships of receptor activator of nuclear factor-kappa B ligand (RANKL) to baseline BMD | baseline visit
The relationships of receptor activator of nuclear factor-kappa B ligand (RANKL) to baseline volumetric BMD | baseline visit
Dose limiting toxicities (DLTs), including hypocalcemia | 3 days, 1 week, 2, week, month 3,4,5,6 after each dose; or any other visits.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Imel, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States